CLINICAL TRIAL: NCT03556618
Title: A Pilot Trial of a Network Intervention for Youth After Incarceration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not feasible to study the WPC intervention as a clinical trial due to disruptions caused by COVID-19.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Elizabeth Barnert, MD, MPH, MS, Principal Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K23DA045747-01 (NIH)
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Youth Incarceration; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Person Care (WPC) Reentry Program - Post-Release (Experimental): In partnership with LA County Health Agency, Dr. Barnert is adapting the successful Transitions Clinic model developed for reentry adults, to assist recently incarcerated transition age youth link to needed health services and reduce substance use disorder relapse and recidivism. This adaption is informed by Dr. Barnert's prior research on the needs of incarcerated adolescents. The intervention, called the "Whole Person Care (WPC) Reentry Program" will consist of community health workers (i.e. network coaches) who are formerly incarcerated and formally trained in care coordination and social network coaching, who interact with justice-involved transition age youth pre- and post-release to increase youths' engagement in community SUD and mental health services. Participants in this branch will include youth exiting the adult justice system (ages 18-24) who receive PRE- and POST-release WPC services.
  Interventions: Behavioral: Whole Person Care (WPC) Reentry Program - Pre & Post Release services
- Control (No Intervention): Participants in the control arm will receive PRE-release services only from Whole Person Care. They will not receive the POST-release WPC community health worker intervention. Participants in this branch will include youth exiting the adult jail system (ages 18-24).

INTERVENTIONS:
Behavioral: Whole Person Care (WPC) Reentry Program - Pre & Post Release services — Social network intervention to provide care coordination and social support during youth reentry before release and post-release from jail.
  Arms: Whole Person Care (WPC) Reentry Program - Post-Release

SUMMARY:
A vicious cycle exists between adolescent substance use disorders and youth incarceration. Re-wiring adolescent social networks during community reentry after incarceration can potentially break the cycle of adolescent substance use and youth incarceration. Social networks influence adolescent substance use and delinquent behavior, yet little is known about how to intervene on social networks to improve health. Community reentry is a key opportunity to re-set youths' social networks and re-direct high-risk youth toward a healthier, more supportive network that can foster drug abstinence and reduce recidivism. The investigators hypothesize that an adult who has successfully navigated reentry can guide youth to rewire their social network by encouraging pro-social relationships, troubleshooting basic barriers to healthcare and social services, and helping create linkages to substance use and mental health treatment services. The goal of this study is to measure the impact of a pilot intervention to address two key barriers to accessing behavioral health treatment among recently incarcerated youth: poor care coordination and need for more positive support from the social network. The proposed study intervention, the Whole Person Care (WPC) Reentry Program, is based on the successful adult Transitions Clinic model, and is being adapted for delivery to transition age youth (TAY) by community partners in the Los Angeles County justice system. WPC community health workers (coaches) will provide recently released inmates a formerly incarcerated adult role model who provides care coordination and social support to facilitate access to needed health services, and who actively intervenes to guide TAY youth toward pro-social peers and adults. The investigators propose a pilot longitudinal study of WPC, using a community-partnered participatory research approach. The primary outcome will be reductions in adolescent substance use in response to the intervention (Aim 1). Secondary outcomes will test whether the intervention increases receipt of behavioral health services, decreases recidivism and mental health symptoms, and improves school and work engagement (Aim 2). Finally, the investigators will examine social networks as a potential mechanism by measuring whether youth receiving the intervention report healthier social networks (lower proportion of peers engaging in risky behaviors and a higher number of supportive adults) than control youth (Aim 3).

DETAILED DESCRIPTION:
A vicious cycle exists between adolescent substance use disorders (SUD) and youth incarceration. Untreated SUD, often comorbid with mental health problems, contribute substantially to youth incarceration. Among 51,000 US youth detained annually, 50-88% have SUD. Incarceration itself can exacerbate existing mental health disorders and contribute to future substance use. Following incarceration, reentry back into the community of peers and adults is a challenging juncture and a high risk period for re-engaging in substance use. Finally, relapse on substance use leads to recidivism. Within 3 years of release, 75% of adolescents are re-arrested, with highest risk among youth with SUD.

Re-wiring adolescent social networks during reentry can potentially break the vicious cycle of adolescent substance use and youth incarceration. Social networks powerfully influence adolescent substance use and delinquent behavior, yet little is known about how to intervene on social networks to improve health. In the investigators prior research, the investigators found that incarcerated youth value relationships with supportive adults and peers who can help them succeed in school and stay out of trouble. Most express plans to "stay clean" from drugs and stay away from peers who encourage substance use and delinquent behaviors. Yet, during reentry, many youth re-engage with their previous network of risky peers. Why? The investigators have found that upon reentry, youth who lack sufficient social supports and positive role models default back to previous risky social networks, reinforcing further substance use and other risky behaviors. Community reentry is a key opportunity to re-set social networks and re-direct high-risk youth toward a healthier network that can foster drug abstinence and reduce recidivism. Having an available and supportive adult role model can be transformative for youth after incarceration. The investigators hypothesize that an adult who has successfully navigated reentry can actively guide youth to re-wire their social network by encouraging pro-social relationships, troubleshooting basic barriers to healthcare and social services, and creating linkages to SUD and mental health services, to disrupt the viscous cycle.

This community-partnered study seeks to measure the impact of an innovative pilot intervention, the Whole Person Care (WPC) Reentry Program, a network community health worker (i.e. coach) intervention that addresses two key challenges for recently incarcerated transition age youth (TAY): poor care coordination in the "behavioral health cascade" and need for more positive support from the social network. Los Angeles (LA) County has the largest adult and juvenile justice systems in the US and has implemented the WPC Reentry Program to enhance linkages to community behavioral health services. WPC is based on the successful Transitions Clinic model, an intervention with demonstrated efficacy in linking recently incarcerated adults to needed healthcare and improving health outcomes. The model has yet to be implemented for reentry TAY, but has the potential to be transformative at the critical developmental stage of adolescence, when peer social networks are highly dynamic and youth behaviors can affect lifelong trajectories. WPC community health workers will receive formalized training modeled after the adult Transitions Clinic approach and will serve as a formerly incarcerated adult role model who provides care coordination and social support to facilitate access to needed behavioral health services. Tailored for reentry youth, WPC will also include a social network component whereby coaches are trained to actively guide youth toward pro-social peers and adults. Dr. Barnert has been working closely with LA County and this study capitalizes on a unique opportunity to rigorously study WPC. The investigators hypothesize that (1) WPC will reduce adolescent SUD and recidivism and (2) WPC will demonstrate positive associations with other key markers of healthy reentry (e.g., improved mental health). The investigators further hypothesize that shifts towards healthier social networks will mediate these relationships, a potential mechanism the investigators will test.

The investigators propose a pilot longitudinal study of WPC, using a community-partnered, participatory research approach. Specific aims are to:

1. Measure the impact of the WPC network coach intervention targeting recently incarcerated youth on decreasing rates of 30-day use and risky use of marijuana, alcohol, and other drug use.
2. Test whether the WPC network coach intervention decreases recidivism, increases receipt of behavioral health services, improves mental health, and enhances school and work engagement.
3. Examine whether recently incarcerated youth receiving the WPC intervention report healthier social networks (lower proportion of peers engaging in risky behaviors and a higher number of supportive adults) than those not receiving the intervention.

ELIGIBILITY:
Inclusion criteria for youth exiting the adult justice system:

* Recipient of WPC pre-release reentry intervention (determined by Los Angeles County)
* Ages 18-24
* Fluent in English or Spanish

Exclusion criteria for youth exiting the adult justice system:

* Not receiving WPC pre-release reentry intervention (determined by Los Angeles County)
* Severe cognitive delay
* Unable to complete surveys in English or Spanish

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth S Barnert, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Los Angeles County Jails, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available to other researchers. The participants, justice-involved youth, are a vulnerable population and we do not currently have permission to share their IPD.

RESULTS

PARTICIPANT FLOW:
Groups:
- Whole Person Care (WPC) Reentry Program - Post-Release: Participants in this branch will include youth exiting the adult justice system (ages 18-24) who receive PRE- and POST-release WPC services.
Period: Overall Study
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Started | 0 | 19
Completed | 0 | 5
Not Completed | 0 | 14

BASELINE CHARACTERISTICS:
Population: 0 participants received the post-release WPC reentry intervention.
Groups:
- Whole Person Care (WPC) Reentry Program: In partnership with LA County Health Agency, Dr. Barnert is adapting the successful Transitions Clinic model developed for reentry adults, to assist recently incarcerated transition age youth link to needed health services and reduce substance use disorder relapse and recidivism. This adaption is informed by Dr. Barnert's prior research on the needs of incarcerated adolescents. The intervention, called the "Whole Person Care (WPC) Reentry Program" will consist of community health workers (i.e. network coaches) who are formerly incarcerated and formally trained in care coordination and social network coaching, who interact with justice-involved transition age youth pre- and post-release to increase youths' engagement in community SUD and mental health services. Participants in this branch will include youth exiting the adult justice system (ages 18-24).
  Whole Person Care (WPC) Reentry Program: Social network intervention to provide care coordination and social support during youth reentry.
- Control: Participants in the control arm will receive usual care reentry healthcare planning post-release, including correctional health provider and court-referred SUD and mental health treatment recommendations, medication prescriptions, written instructions for reinstating Medicaid, and written health discharge summaries. Participants in this branch will include youth exiting the adult justice system (ages 18-24) and youth exiting the juvenile justice system (ages 16-18).
- Total: Total of all reporting groups
Arm/Group | Whole Person Care (WPC) Reentry Program | Control | Total
Number analyzed (Participants) | 0 | 19 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 19 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 22 [18 to 24] | 22 [18 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 19 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 9 | 9
  Not Hispanic or Latino | 0 | 10 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 7 | 7
  White | 0 | 10 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 19 | 19
30-day Marijuana Use [Mean (Standard Deviation); unit: days] |  | 22.9 (13.1) | 22.9 (13.1)
30-day Alcohol Use [Mean (Standard Deviation); unit: days] |  | 13.1 (14.2) | 13.1 (14.2)
Mental Health [Count of Participants; unit: Participants] — self reported mental health diagnosis
  Participants |  | 7 | 7
Arrest History [Mean (Standard Deviation); unit: arrests] |  | 10.4 (9.8) | 10.4 (9.8)
Substance Use Disorder [Count of Participants; unit: Participants] |  | 13 | 13
Medications [Count of Participants; unit: Participants] |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Past-month (30-day) Marijuana Use
Description: Self-reported frequency of past-month (30-day) marijuana use
Time Frame: 3 months post-release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
days |  | 7.4 (10.9)

2. Primary Outcome: Frequency of Past-month (30-day) Alcohol Use
Description: Self-reported frequency of past-month (30-day) alcohol use
Time Frame: 3 months post-release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
days |  | 2 (2.8)

3. Secondary Outcome: Frequency of Past-month (30-day) Marijuana Use
Description: Self-reported frequency of past-month (30-day) marijuana use
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
days |  | 10 (11.8)

4. Secondary Outcome: Frequency of Past-month (30-day) Alcohol Use
Description: Self-reported frequency of past-month (30-day) alcohol use
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
days |  | 2 (2.8)

5. Secondary Outcome: Recidivism
Description: Re-arrest since release (self-report and administrative/probation data)
Time Frame: 3 months post-release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: arrests
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
arrests |  | 0.6 (1.1)

6. Secondary Outcome: Recidivism
Description: Re-arrest since last survey (self-report and administrative/probation data)
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: arrests
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
arrests |  | 0.2 (0.4)

7. Secondary Outcome: Receipt of Behavioral Health Services
Description: receipt of behavioral since release (self-report and verified by administrative/probation data)
Time Frame: 3 months post-release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 7

8. Secondary Outcome: Receipt of Behavioral Health Services
Description: receipt of behavioral since last survey (self-report and verified by administrative/probation data)
Time Frame: 9 months post-release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 5

9. Secondary Outcome: Mental Health
Description: self-reported presence of diagnosis of a mental health disorder (will be verified by administrative/probation data)
Time Frame: 3 months post release
Population: No participants were in the treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants | 0 | 2

10. Secondary Outcome: Mental Health
Description: self-reported presence of diagnosis of a mental health disorder at follow-up (will be verified by administrative/probation data)
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 1

11. Secondary Outcome: Substance Use Disorders
Description: self-reported presence or diagnosis of substance use disorder at follow-up (will be verified by administrative/probation data)
Time Frame: 3 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 1

12. Secondary Outcome: Substance Use Disorders
Description: as for outcome 11
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 0

13. Secondary Outcome: Medications
Description: self-reported medication or prescription at follow-up (will be verified by administrative/probation data)
Time Frame: 3 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 4

14. Secondary Outcome: Medications
Description: self-reported medication or prescription at follow-up (will be verified by administrative/probation data)
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 1

15. Secondary Outcome: Delinquency
Description: number of arrest since release (will be verified by administrative/probation data)
Time Frame: 3 months post release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: arrests
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
arrests |  | 0.6 (1.1)

16. Secondary Outcome: Delinquency
Description: number of arrest since last survey (will be verified by administrative/probation data)
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Mean (Standard Deviation); unit: arrests
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
arrests |  | 0.2 (0.4)

17. Secondary Outcome: Attitudes Towards WPC Reentry Intervention (WPC Reentry Participant Response Tool)
Description: Liked intervention; recommend to a friend. Assessed via WPC Reentry Participant Response Tool. Includes 3 items, assessed via 7-point Likert scale.
Time Frame: 3 months post release
Population: No participants were in the intervention arm of the study. This question asked about the intervention and was therefore skipped for participants in the control arm
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Attitudes Towards WPC Reentry Intervention (WPC Reentry Participant Response Tool)
Description: as for outcome 17
Time Frame: 9 months post release
Population: as for outcome 17
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Psychiatric Hospitalizations
Description: psychiatric hospitalizations since release (self-report and health records data)
Time Frame: 3 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 1

20. Secondary Outcome: Psychiatric Hospitalizations
Description: psychiatric hospitalizations since last survey (self-report and health records data)
Time Frame: 9 months post release
Population: No participants were in the intervention arm of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Person Care (WPC) Reentry Program - Post-Release | Control
Number analyzed (Participants) | 0 | 19
Participants |  | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: The number at risk for adverse events in the WPC arm is 0 because no participants enrolled in WPC post-release. Thus, 0 participants were in the intervention arm of the study, and no intervention-arm participants were at-risk of adverse events
Arm/Group | Whole Person Care (WPC) Reentry Program | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/19
Other Adverse Events (participants affected / at risk) | 0/0 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03556618/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03556618/SAP_001.pdf
  • Informed Consent Form (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03556618/ICF_002.pdf